CLINICAL TRIAL: NCT00704275
Title: Comparison of Efficacy, Safety and Anti-Inflammatory Effect Between Topical 0.05%Cyclosporine A Emulsion and REFRESH® in Patients With Moderate to Severe Dry Eyes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Vilavun Puangsricharern/Ass. Prof in Ophthalmology, Department of Ophthalmology, Faculty of Medicine, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 391/48
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Last update posted 2008-06-24 (Estimated); Status verified 2008-06

CONDITIONS: Dry Eye
Keywords: dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 0.05% cyclosporin
  Interventions: Drug: 0.05% cyclosporin eye drop
- B (Active Comparator): Refresh
  Interventions: Drug: 0.05% cyclosporin eye drop

INTERVENTIONS:
Drug: 0.05% cyclosporin eye drop — bid dosage for 4 months

SUMMARY:
To compare the efficacy, safety and tolerability of 0.05% topical cyclosporin eye drop to Refresh in moderate to severe dry eye patients. Null hypothesis is: there is no difference between these two groups.

DETAILED DESCRIPTION:
Inclusion criteria:

1. Participants are moderate to severe dry eye patients aged more than 18 years of age
2. Oxford staining scores of more than five.
3. OSDI scores of more than 0.1

Outcome measurements:

Main parameter is staining score (corneal + conjunctival) Other parameter is OSDI score, symptom of ocular surface discomfort score, number of daily artificial tear needed, TBUT, Schirmer I score, cytokines level & markers Safety parameters: VA, IOP, cyclosporin level

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe dry eye

Exclusion Criteria:

* lid anomaly, previous CsA use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-07 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Corneal and conjunctival staining score | 1 year

SECONDARY OUTCOMES:
Schirmer 1 score | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- OPD Chulalongkorn University Hospital, Bangkok, Thailand